CLINICAL TRIAL: NCT06261528
Title: A Phase I Study of Circadian Focused Light Therapy for Fatigue Reduction in Progressive Multiple Sclerosis (NO-FATIGUE)
Brief Title: Study of Circadian Focused Light Therapy in Progressive Multiple Sclerosis
Acronym: NO-FATIGUE
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Sguigna, Assistant Professor - Department of Neurology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1289
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Fatigue; Sleepiness; Circadian
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Fatigue; Sleepiness | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: This will be an open label, single arm, single center phase 1 research study designed to generate safety data, biomarker data, and preliminary efficacy data to reduce fatigue in patients with progressive MS, to include PPMS and SPMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Circadian Focused Light Therapy for Fatigue Reduction in Progressive Multiple Sclerosis (NO-FATIGUE) (Experimental): This will be an open label, single arm, single center phase 1 research study designed to generate safety data, biomarker data, and preliminary efficacy data to reduce fatigue in patients with progressive MS, to include PPMS and SPMS
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — Light therapy aimed at alleviating fatigue through circadian rhythm synchronization

SUMMARY:
The study is being done to determine if treatment with a novel form of light therapy is tolerated in patients with progressive multiple sclerosis. The goal of this trial to establish the safety profile of this light therapy while generating data on its impact on fatigue, as well as its mechanism of action. Fatigue is often a complex symptom in multiple sclerosis, without any FDA-approved direct therapy. Fatigue is traditionally treated with symptom management through a multidisciplinary team.

DETAILED DESCRIPTION:
This will be an open label, single arm, single center, phase 1 research study designed to determinate the safety and mechanism of action of targeted light therapy as a treatment for fatigue in people with progressive multiple sclerosis (PMS).

Participants will undergo a 2-week screening that includes an at home sleep monitor, saliva collection, and completion of surveys. Once screening is complete, participants will complete a light therapy program that will require visits to UT Southwestern Medical Center each day for 3 days, and then every 2-3 weeks for three visits, for a total of 7 visits. Each visit will take about 3 hours. Participants will also be asked to collect saliva, wear the home sleep monitor, and complete surveys. The total study duration is about 2.5 months.

The risks of this study include the possibility of eye irritation during the light therapy, and loss of confidentiality.

The primary outcome will be the treatment emergent adverse events. There is a number of exploratory efficacy and mechanism of action outcomes for future study design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of PPMS or SPMS according to the 2017, or 2010 Revised McDonald Criteria
* In the opinion of the investigator, able to complete study procedures
* Epworth Sleepiness Scale (ESS) ≥ 9
* Must be on a stable dose of an FDA-approved disease modifying therapy for at least 3 months prior to screening
* Pharmacological and non-pharmacological mood and fatigue treatments must be stable for the previous three months prior to screening and must have intent to keep these stable for the duration of study treatment

Exclusion Criteria:

* Sleep onset latency under 15 minutes
* Pharmacological and non-pharmacological mood and fatigue treatments changes within the previous three months prior to screening
* Based on the Investigator's judgement, patients with a history of significant other medical condition that may interfere with the conduct of the study, or interpretation of the study results
* History of any clinically significant abnormality in hematology, blood chemistry, or examination not resolved by the baseline visit which according to the investigator can interfere with study participation
* Positive drug screen for cocaine, or phencyclidine, or known alcohol abuse within 30 days of the trial
* Females who are pregnant, have a provided recent positive pregnancy test, are nursing, or who plan to get pregnant during the course of this clinical trial
* Patient taking melatonin analogues without appropriate washout, defined as five half-lives of the medication, or within 14 days of screening, whichever is longer
* No new or adjusted prescription medication within 14 days of the baseline
* An investigator verified MS relapse within the previous year
* Presence of a gadolinium-enhancing demyelinating lesion within the last year
* Optic neuritis within the previous 3 months
* Sleep schedule changes as required by employment (night shifts)
* Travel across two time zones within 3 months of study screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | 2.5 months
  The primary objective is to characterize treatment emergent adverse events (TEAEs) following light therapy targeting circadian rhythm synchronization. Data will be summarized descriptively as incidence/prevalence relative to the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sguigna, MD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that supports a publication as reported in the article after deidentification will be available to qualified investigators with reasonable requests.
Supporting Information: Study Protocol
Time Frame: The data will be available within two years of publication of the results of the trial by qualified investigators for a defined period of time. This data will be available through institutional mechanisms.